CLINICAL TRIAL: NCT04209894
Title: Detection of Subclinical Enthesitis by Ultrasonography in Psoriasis Patients With Psoriasis and Controls: by Ultrasonography; Incidence of Psoriatic Arthritis During Within One 1 Year
Brief Title: Detection of Subclinical Enthesitis by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Karamanlıoğlu, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: karamanlioglu.duygu
Record Dates: First submitted 2019-12-14; First posted 2019-12-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Enthesitis
Keywords: subclinical enthesitis; psoriasis; ultrasound; psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriasis: They will undergo dermatological assessment and a blinded ultrasound (US) evaluation.
  Interventions: Diagnostic Test: Ultrasound
- Control: They will also undergo dermatological assessment and a blinded ultrasound (US) evaluation.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Evaluation consisted of the detection of grey scale (GS) enthesitis and Power Doppler signal in enthesis areas of participants. The Madrid Sonography Enthesitis Index (MASEI) scoring system was used to quantify the extent of sonographic entheseal abnormalities

SUMMARY:
Detection of subclinical enthesitis by ultrasonography

DETAILED DESCRIPTION:
A total of 30 patients with psoriasis and 30 age-matched healthy controls, all without musculoskeletal diseases, will be recruited. They will undergo dermatological assessment and a blinded ultrasound (US) evaluation. Clinical assessment included demographics, severity of psoriasis and musculoskeletal clinical examination. Evaluation consisted of the detection of grey scale (GS) enthesitis and Power Doppler signal in enthesis areas. The Madrid Sonography Enthesitis Index (MASEI) scoring system was used to quantify the extent of sonographic entheseal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18years
* Patients with psoriasis without musculoskeletal symptoms
* Healthy controls
* No joint involvement and no clinical symptoms and signs of enthesitis and synovitis

Exclusion Criteria:

* Have history of gout or arthritis or peripheral neurological disease of lower extremity.
* Have history of trauma and intensive sport activity in last 2 weeks.
* Have received any systemic therapy (i.e. DMARD, NSAIDs, corticosteroids, immunosuppressants, retinoids or biological agents) in 3 months
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both patients with psoriasis and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Detection of Subclinical Enthesitis by Ultrasonography in Psoriasis Patients with Psoriasis and Controls: by Ultrasonography; Incidence of Psoriatic Arthritis During Within One 1 Year | 1 year.
  Incidence of subclinical enthesitis,To investigate the incidence of subclinical enthesitis in patients with psoriasis

SECONDARY OUTCOMES:
Number of participants with Risk factors of subclinical enthesitis | 1 year
  To find out predictor factors of subclinical enthesitis in patients with psoriasis. To assess increase in enthesis area and PsA incidence, and show a possible relationship with baseline findings in a prospective 1-year follow-up of patients with PsO.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Silte Karamanlioglu, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital; Feyza Unlu Ozkan, Prof., Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Eylem Ceren Arikan, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Betül Zehra Pirdal, MD, Study Chair — Istanbul Sultangazi District Health Directorate; Gulcan Ozturk, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Ilknur Aktas, Prof, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No